CLINICAL TRIAL: NCT07203742
Title: The Effect of Mandala on Anxiety and Fear Levels in Children With Leukemia Before Intrathecal Chemotherapy Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, SEDA ARDAHAN SEVGİLİ, Asst. Professor, Ege University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 25-9.1T/59
Record Dates: First submitted 2025-09-23; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Acute Lymphoblastic Leukemia; Childhood Acute Leukemia; Acute Myeloblastic Leukaemia
Keywords: intrathechal chemotherapy treatment; anxiety; fear; mandala; nursing
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mandala painting (Experimental)
  Interventions: Other: mandala painting
- control (No Intervention)

INTERVENTIONS:
Other: mandala painting — After the child and parent agree to participate in the study and the child indicates that they wish to do the mandala exercise, the child will be seated in a comfortable position to paint. Thirty minutes before the start of the intrathecal chemotherapy procedure (children who will receive intrathecal chemotherapy at the clinic are identified and scheduled the day before), the child, their parent, and a nurse independent of the study will be assessed using the "Child Anxiety Scale-State (ÇAS-D)" and the "Child Fear Scale." The mandala coloring activity will then continue until the child wishes to stop (the activity will be ensured to last at least 30 minutes). When the child is called to the procedure room for intrathecal chemotherapy, the scale assessments will be repeated. Thirty minutes after the intrathecal chemotherapy procedure is completed and the child has emerged from the effects of general anesthesia, the scales will be reassessed and recorded by the same i
  Arms: mandala painting

SUMMARY:
This study aims to examine the effect of mandala coloring activity, administered before intrathecal chemotherapy treatment in children with leukemia, on pre-procedure anxiety and fear in children. The main question this study aims to answer is:

Does mandala coloring administered before intrathecal chemotherapy treatment reduce pre-procedure anxiety and fear in children with leukemia?

Descriptive demographic data will be collected from the children who will be given mandalas. Data will be collected using an Anxiety Scale and a Fear Scale.

DETAILED DESCRIPTION:
Acute leukemia, the most common cancer in childhood (32% in girls and boys aged 0-14), is characterized by the uncontrolled and abnormal proliferation of leukocytes in the bone marrow, where blood cells are produced. Chemotherapy agents are used in its treatment. Subsequently, intrathecal chemotherapy is administered according to the child's risk group and protocol. Intrathecal chemotherapy options include intrathecal methotrexate or a combination of intrathecal methotrexate with cytarabine and hydrocortisone. Numerous complications associated with chemotherapy may occur. These complications include fatigue, nausea and vomiting, hair loss, pancytopenia, mucositis, diarrhea, and constipation. In addition, psychological side effects such as depression, anxiety, fear, and insomnia are also frequently seen in children. Non-pharmacological methods are available for managing psychological side effects in individuals diagnosed with leukemia. These methods include psychoeducation, cognitive-behavioral therapy, art therapy, supportive psychotherapy, relaxation, and distraction techniques. In addition to these methods, mandala coloring, which can be used in many different situations, is also available. This study aims to investigate the effect of mandala coloring activity on anxiety and fear levels in children with leukemia before intrathecal treatment. The study will be conducted at the Pediatric Hematology Clinic of Ege University Faculty of Medicine Children's Hospital with a total of 60 children aged 4-12 years who are scheduled for intrathecal treatment. Children aged 4-12 years who meet the inclusion criteria and who will receive intrathecal chemotherapy due to leukemia treatment will be included in the study. The "Unmatched Control Group Model" will be used in the study, and randomization will not be performed. In this design, the intervention and control groups are planned to consist of participants with similar characteristics. To prevent/minimize interaction between groups, the control group data will be collected first. After the control group data is collected, the intervention group data will be collected. Data collection and the intervention will be carried out after the children are assigned to their groups. The SPSS 26.0 software package will be used to analyze the data obtained after the study. Frequency and percentage distributions will be used to check the distribution of participants' demographic characteristics and the normality of the data. Advanced analyses will then be performed.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be between 4 and 12 years of age.
* The patient must be hospitalized and followed up at the Pediatric Hematology Clinic.
* The patient must only be receiving leukemia treatment.
* The patient must not have any other chronic diseases.
* The patient must not have any systemic infections.
* The patient has received at least two courses of intrathecal chemotherapy treatment
* The patient does not have a diagnosis of psychological/mental symptoms as a side effect of chemotherapy treatment
* Intrathecal treatment will be administered to the patient in accordance with the chemotherapy protocol
* The patient and the caregiver parent are volunteers
* The caregiver parent speaks Turkish and is open to communication.

Exclusion Criteria:

* Cases that do not meet the inclusion criteria will be excluded from the study.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-09-29 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Fear of intrathecal chemotherapy | From enrollment to 30 minutes after intrathecal chemotherapy
  The fear that children will experience due to intrathecal chemotherapy will be collected using the "Children's Fear Scale".
Anxiety of intrathecal chemotherapy | From enrollment to 30 minutes after intrathecal chemotherapy
  The fear that children will experience due to intrathecal chemotherapy will be collected using the "Children's Anxiety Scale".

CONTACTS AND LOCATIONS:
Overall Officials: Seda Ardahan Sevgili, Ph.D., Principal Investigator — Ege University

IPD SHARING:
Plan to Share IPD: No